CLINICAL TRIAL: NCT01081327
Title: Observational Record Linkage Study Investigating Incidence of Adverse Events in Patients Anti-coagulated for Lone Atrial Fibrillation.
Brief Title: Warfarin - How Good Are we at Maintaining Target Range ?
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Sponsor
Other Study IDs: ELD007
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2010-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Warfarin; Safety
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving Warfarin

SUMMARY:
Patients with atrial fibrillation are often anticoagulated with Warfarin. Warfarin has a narrow therapeutic window requiring frequent monitoring. This study aims to investigate the incidence of adverse events in the "real world" for patients receiving Warfarin for lone atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Prescription for Warfarin
* Atrial Fibrillation

Exclusion Criteria:

* Other conditions associated with increased risk of embolisation e.g. rheumatic valve disease, atrial mixoma.
* Conditions with increased risk of bleeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving Warfarin for lone atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2010-03; Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Bleeding Complication | 10 years
  Any bleeding event requiring hospitalisation and / or blood transfusion. Any death attributable to bleeding i.e. Intracerebral bleed.
Cardiovascular outcome | 10 years
  Ischaemic event e.g. Cerebral infarction / Myocardial infarction / death attributed to ischaemic event

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Cardiovascular and Lung Biology, Univeristy of Dundee, Dundee, United Kingdom